CLINICAL TRIAL: NCT01989182
Title: The Spiration Valve System for the Treatment of Severe Emphysema
Acronym: REACH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Olympus Corporation of the Americas (Industry)
Collaborators: Olympus Corporation (Industry); Tigermed Consulting Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TG1226SVS
Record Dates: First submitted 2013-11-06; First posted 2013-11-20 (Estimated); Last update posted 2018-02-14 (Actual); Status verified 2018-02

CONDITIONS: Empyhsema; Pulmonary Disease, Chronic Obstructive
Keywords: Endobronchial Valves; Intrabronchial Valves; Bronchial Valve; Chronic Obstructive Pulmonary Disease; COPD; Pulmonary Disease, Chronic Obstructive; Bronchoscopic Lung Volume Reduction; BLVR; TLVR; Emphysema; Pulmonary Emphysema; Pathologic Process; Lung Diseases; Respiratory Tract Disease; China; Spiration Valve System (SVS)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema; Pulmonary Emphysema; Pathologic Processes; Lung Diseases; Respiratory Tract Diseases | interventions — Practice Management, Medical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment with Spiration Valve System (Experimental): Subjects assigned to the treatment group will undergo a bronchoscopic procedure to have valves placed in the most diseased lobe of the lung to occlude all segments of the lobe. Subjects assigned to this group will also receive medical management.
  Interventions: Device: Spiration Valve System; Other: Medical Management
- Medical Management (Active Comparator): The control group for this study will receive medical management. This medical management group will be evaluated and followed in the same manner as the treatment group, but without having a bronchoscopic procedure.
  Interventions: Other: Medical Management

INTERVENTIONS:
Device: Spiration Valve System
  Arms: Treatment with Spiration Valve System
Other: Medical Management

SUMMARY:
This is a multicenter, prospective, randomized, controlled study being conducted in China to evaluate improvement of lung function after treatment with the Spiration Valve System as compared to medical management in the control group. The control group will be evaluated in the same manner as the treatment group.

The Spiration Valve is a small, umbrella-shaped, one-way valve that is placed inside the airways of one lung. It is used to redirect air from the less healthy to the more healthy parts of the lung. This helps to reduce over-inflation and may improve overall lung function and quality of life for people living with emphysema.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has severe emphysema and high heterogeneity by visual assessment defined as:

   * a target lobe with ≥ 40% emphysema involvement and
   * ≥ 15% difference with the ipsilateral lobe.
2. The target lobe and ipsilateral lobe will be separated with an intact fissure. An intact fissure will be estimated visually to be ≥90% complete after viewing the HRCT in 3 dimensions.
3. Patient has received optimal medical management and it has been stable for 6 weeks prior to baseline testing. If pulmonary rehabilitation has been recent, it will be completed at least 3 months prior to baseline testing.
4. Patient must be able to demonstrate physical ability to participate in the study by performing a 6-minute walk distance of ≥ 140 m.
5. Patient has abstained from cigarette smoking for 4 months and is willing to abstain throughout the study.
6. Severe dyspnea defined as a mMRC ≥ 2.
7. Patient's obstructive disease is severe as defined by:

   * FEV1 ≤ 45% of predicted
8. Patient's hyperinflation is defined by:

   * TLC ≥ 100% of predicted
   * RV ≥ 150% of predicted
9. Patient is willing to participate in a study, complete the required follow-up visits, and maintain consistent nutrition and exercise habits during the study period.
10. Investigator has confirmed that medical management is within standard of care and patient has been stable and without a COPD exacerbation for 6 weeks or more.

Exclusion Criteria:

1. Patient has severe gas exchange abnormalities as defined by:

   * PCO2 > 50 mm Hg (6.6 kPa), or
   * PaO2 < 45 mm Hg (6.0 kPa) on room air
2. Patient has a BMI < 15 kg/m2 or > 35 kg/m2
3. Patient is unable to provide informed consent.
4. Patient is not an appropriate candidate for or is unable to tolerate, flexible bronchoscopy procedures.
5. Patient has dysrhythmia or cardiovascular disease that poses a risk during exercise.
6. Patient has history of 4 or more hospitalizations for COPD exacerbation or respiratory infections in the past year or has had a COPD exacerbation in the 3 months prior to baseline testing.
7. Patient has bronchitis with sputum production > 60 ml per day.
8. Patient has an active asthma component to their disease or requires more than 15 mg of prednisone daily (20 mg prednisolone).
9. Patient has giant bulla (> 1/3 volume in either lung).
10. Patient has severe pulmonary hypertension based upon clinical evaluation.
11. A patient with a malignant condition and/or a life threatening disease (other than COPD) that would likely affect the completion of the study
12. Patient has any disease or condition that interferes with completion of initial or follow-up assessments of the effectiveness endpoints. This would include neurological or musculoskeletal conditions that may interfere with testing.
13. Patient has had prior lung volume reduction surgery or major lung procedures (lobectomy or greater).
14. Patient has a lung nodule anticipated to require evaluation or intervention during the 3 month study period.
15. Patient has demonstrated unwillingness or inability to complete screening or baseline data collection procedures.
16. Patient has a diffuse emphysema pattern, diffuse pulmonary fibrosis, or pulmonary tuberculosis (active, extensive, or with adhesive pleural incrassation).
17. Patient is classified as ASA Class greater than P4 including presence of co-morbidity that could significantly increase the risk of a bronchoscopy procedure.
18. Patient participated in a study of an investigational drug or device within the past 30 days prior to participation in this study, or is currently participating in another clinical study.
19. Female patient of childbearing potential has a positive result from a pregnancy test required during the 7 days prior to the procedure.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2013-11-08 (Actual); Primary Completion 2016-05-18 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Difference between treatment and control groups in the mean change in forced expiratory volume in one second (FEV1) | Baseline and 3 Months

SECONDARY OUTCOMES:
Incidence of device-related serious adverse events | Baseline and 3 Months
Difference between responder rates in the treatment and control groups, with a responder defined as ≥ 15% improvement in FEV1 | Baseline and 3 Months
Target lobe volume reduction as measured by QCT | Baseline and 3 Months
Health Status as measured by St. George's Respiratory Questionnaire (SGRQ) and COPD Assessment Test (CAT) | Baseline and 3 Months
Dyspnea as measured by Modified Medical Research Council Questionnaire (mMRC) | Baseline and 3 Months
Exercise capacity as measured by Six Minute Walk Test (6MWT) | Baseline and 3 Months
Hyperinflation as measured by Residual Volume (RV) | Baseline and 3 Months

CONTACTS AND LOCATIONS:
Overall Officials: Nanshan Zhong, MD, Principal Investigator — The First Affiliated Hospital of Guangzhou Medical University
Locations (12):
- China (12):
  - Guangdong General Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - Tangdu Hospital the Second Teaching Hospital of the Fourth Military Medical University, Xi'an, Shaanxi
  - The First Affiliated Hospital of Wenzhou Medical College, Wenzhou, Zhejiang
  - Peking University First Hospital, Beijing
  - The General Hospital of Chinese People's Liberation Army (301), Beijing
  - The Second Affiliated Hospital ZheJiang University School of Medicine, Hangzhou
  - Shanghai Chest Hospital, Shanghai
  - Shanghai Tenth People's Hospital, Shanghai
  - Zhongshan Hospital Fudan University, Shanghai